CLINICAL TRIAL: NCT06021951
Title: An Open-Label Postmarking Milk-Only Lactation Study to Evaluate the Concentration of Bempedoic Acid and Bempedoic Acid and Ezetimibe in the Breast Milk of Healthy Lactating Women Administered Therapeutic Doses of Bempedoic Acid or Bempedoic Acid/Ezetimibe Fixed Combination Drug Product (FCDP)
Brief Title: Milk-Only Lactation Study to Evaluate the Concentration of Bempedoic Acid and Bempedoic Acid/Ezetimibe Fixed Combination Drug Product (FCDP) in the Breast Milk of Healthy Lactating Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1002FDC-075
Record Dates: First submitted 2023-08-27; First posted 2023-09-01 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-05

CONDITIONS: Healthy Lactating Women
Keywords: Bempedoic acid; Ezetimibe; Bempedoic acid and ezetimibe; Breast Milk
MeSH Terms: interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bempedoic acid (Experimental)
  Interventions: Drug: Bempedoic Acid 180 MG Oral Tablet
- Bempedoic acid/ezetimibe fixed combination drug product (Experimental)
  Interventions: Drug: Bempedoic Acid/Ezetimibe 180 MG-10 MG Oral Tablet

INTERVENTIONS:
Drug: Bempedoic Acid 180 MG Oral Tablet — Bempedoic Acid 180 MG Oral Tablet [Nexletol]
  Other Names: Nexletol
  Arms: Bempedoic acid
Drug: Bempedoic Acid/Ezetimibe 180 MG-10 MG Oral Tablet — Bempedoic Acid/Ezetimibe 180 MG-10 MG Oral Tablet [NEXLIZET]
  Other Names: Nexlizet 180 mg-10 mg
  Arms: Bempedoic acid/ezetimibe fixed combination drug product

SUMMARY:
This study is designed to characterize the excretion of bempedoic acid or bempedoic acid and ezetimibe into mature breast milk of healthy lactating women and assess the exposure to the breast fed infant by estimating the daily infant dosage and the relative infant dose (RID) of bempedoic acid or bempedoic acid and ezetimibe in breast milk after 6 consecutive daily doses of bempedoic acid or bempedoic acid/ezetimibe FCDP.

DETAILED DESCRIPTION:
Post marketing approval commitment for the FDA

ELIGIBILITY:
Inclusion Criteria:

* The subject must be a lactating female who had a normal full-term pregnancy and has been actively breastfeeding or pumping for at least 4 weeks; lactation must be well established per Investigator discretion.
* The subject must be willing to pump regularly during the study to maintain milk supply and discontinue breastfeeding for the entire 13-day Treatment and Washout Periods.
* The subject must not be pregnant.
* The subject must be surgically sterile or willing to use 1 acceptable method of birth control.

Exclusion Criteria:

* Has clinically significant infection (e.g., pneumonia, pyelonephritis) or chronic infection within 30 days prior to enrollment.
* Has evidence of unstable or uncontrolled, clinically significant cardiovascular, central nervous system, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder, including serious allergy, asthma, hypoxemia, hypertension, seizures, or allergic skin rash, that, in the opinion of the Investigator, would confound the study results or compromise subject safety.
* Has estimated glomerular filtration rate (eGFR) <30 mL/min/1.732 using the Modification of Diet in Renal Disease (MDRD) formula.
* Has liver disease or dysfunction characterized by Child-Pugh Class B or Class C.
* History of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.
* Has active psychiatric problems that, in the Investigator's opinion, may interfere with compliance with the study procedures.
* Has history of breast implants, breast augmentation, or breast reduction surgery.
* Has a prior history of difficulty establishing lactation.
* Gastrointestinal conditions or procedures (including weight loss surgery; e.g., Lap-Band® or gastric bypass) that may affect drug absorption.
* Any history of malignancy (with the exception only of basal or squamous cell carcinoma of the skin in individuals that have been cancer free for >5 years).
* History within the last 2 years of drug, alcohol, amphetamine and derivatives, or cocaine abuse.
* Current smoker.
* Blood donation, participation in a multiple blood draw clinical study, major trauma, or surgery with or without blood loss within 30 days prior to enrollment.
* Blood transfusion for any reason within 90 days prior to enrollment.
* Use of any 3-hydroxy-3-methylglutaryl coenzyme A (HMG CoA) reductase inhibitor (statin) concurrently or within 30 days prior to randomization.
* Use of cyclosporine, cholestyramine, probenecid, fibrate drugs, or medications contraindicated during lactation concurrently or within 30 days prior to randomization.
* Concomitant use or use within 30 days prior to randomization of drugs that decrease breast milk production, such as pseudoephedrine.
* Concomitant use or use within 30 days prior to randomization of drugs that increase breast milk production, such as domperidone.
* Use of any experimental or investigational drugs/vaccines concurrently or within 30 days or 5 half-lives of the drug, whichever is longer, prior to screening.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Broestl, MS, Study Director — Esperion Therapeutics, Inc.
Locations (1):
- PPD Development, Las Vegas Research Unit, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 4, open-label study that estimated the daily infant dosage and relative infant dose (RID) for bempedoic acid and bempedoic acid/ezetimibe fixed combination drug product (FCDP) and characterized the excretion of bempedoic acid (ETC-1002), ezetimibe, and metabolites ESP-15228, ETC-1002-glucuronide, and ezetimibe-glucuronide in the mature breast milk of healthy women.
Pre-assignment Details: A total of 16 subjects were enrolled into the study and randomized in a 1:1 ratio to receive bempedoic acid 180 milligrams (mg) or bempedoic acid 180 mg/ezetimibe 10 mg FCDP
Groups:
- Bempedoic Acid: Participants received bempedoic acid 180 mg oral tablet for 6 days
- Bempedoic Acid/Ezetimibe FCDP: Participants received bempedoic acid 180 mg/ezetimibe 10 mg FCDP oral tablets for 6 days
Period: Overall Study
Arm/Group | Bempedoic Acid | Bempedoic Acid/Ezetimibe FCDP
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprised of all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bempedoic Acid | Bempedoic Acid/Ezetimibe FCDP | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.5 (4.17) | 27.1 (4.09) | 30.3 (5.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 8 | 5 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 3 | 4
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Daily Infant Dose
Description: Daily infant dosage of study drug was calculated for Bempedoic Acid arm and FCDP arm respectively from the cumulative amount of study drug (bempedoic acid or bempedoic acid and ezetimibe) excreted in breast milk over 24 hours.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set comprised of all participants in Full Analysis Set who had at least 1 evaluable post-dosing breast milk bempedoic acid pharmacokinetic concentration data point.
Measure: Mean (Standard Deviation); unit: Milligrams per day
Groups:
- Bempedoic Acid: Bempedoic Acid Arm
- Bempedoic Acid (FCDP); Ezetimibe (FCDP): Bempedoic Acid / Ezetimibe FCDP Arm
Arm/Group | Bempedoic Acid | Bempedoic Acid (FCDP) | Ezetimibe (FCDP)
Number analyzed (Participants) | 8 | 8 | 8
Milligrams per day | 0.0331 (0.0210) | 0.0337 (0.0286) | 0.0002 (0.0002)

2. Primary Outcome: Relative Infant Dose (RID)
Description: Relevant Infant Dose (RID) (calculated as the ratio of estimated infant daily dose per kg body weight and maternal daily dose per kg of body weight multiplied by 100) was analyzed for the Bempedoic Acid arm and FCDP arm respectively. Maternal dosage is the ratio of bempedoic acid dose or ezetimibe dose administered daily divided by maternal body weight at baseline.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: Percentage of maternal dose
Arm/Group | Bempedoic Acid | Bempedoic Acid (FCDP) | Ezetimibe (FCDP)
Number analyzed (Participants) | 8 | 8 | 8
Percentage of maternal dose | 0.4790 (0.1962) | 0.4678 (0.2889) | 0.0370 (0.0097)

3. Secondary Outcome: Cumulative Amount of Bempedoic Acid (ETC-1002) and Metabolites (ESP-15228, ETC-1002-Glucuronide) in Breast Milk
Description: Cumulative amount of ETC-1002, ESP-15228, and ETC-1002-glucuronide excreted in breast milk during the 24-hour collection period were analyzed for the Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Nanograms
Groups:
- ETC-1002; ESP-15228; ETC-1002-Glucuronide: Bempedoic Acid Arm
- ETC-1002 (FCDP); ESP-15228 (FCDP); ETC-1002-Glucuronide (FCDP): Bempedoic Acid / Ezetimibe FCDP Arm
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Nanograms | 33120.0 (21034.11) | 14207.4 (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 20690.5 (6554.48) | 33673.4 (28635.66) | 770.0 (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 20709.1 (16012.78)

4. Secondary Outcome: Cumulative Amount of Ezetimibe (EZE) and Metabolite (EZE-Glucuronide) in Breast Milk
Description: Cumulative amount of Ezetimibe, and EZE-glucuronide excreted in breast milk during 24-hour collection period were analyzed (FCDP arm only).
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Mean (Standard Deviation); unit: Nanograms
Groups:
- Ezetimibe; EZE-Glucuronide: Bempedoic Acid / Ezetimibe FCDP Arm
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Nanograms | 182.2 (154.97) | 983.0 (996.16)

5. Secondary Outcome: Maximum Concentrations (Cmax) of Bempedoic Acid and Metabolites in Breast Milk
Description: Cmax of ETC-1002, ESP-15228, and ETC-1002-glucuronide in Breast Milk were analyzed for Bempedoic Acid arm and FCDP arm respectively
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Nanograms per milliliter | 118.15 (38.91) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 73.06 (56.59) | 107.46 (43.19) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 57.29 (56.35)

6. Secondary Outcome: Cmax of Ezetimibe and Metabolite in Breast Milk
Description: Cmax of Ezetimibe, and EZE-glucuronide analyzed in FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 0.63 (44.29) | 2.93 (54.02)

7. Secondary Outcome: Time of Maximum Concentration (Tmax) of Bempedoic Acid and Metabolites in Breast Milk
Description: Tmax of ETC-1002, ESP-15228, and ETC-1002-glucuronide in Breast Milk were analyzed for Bempedoic Acid arm and FCDP arm respectively
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Median (Full Range); unit: Hours
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Hours | 2.94 [2.8 to 6.0] | NA [NA to NA] — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 8.92 [5.7 to 12.0] | 2.93 [2.8 to 8.9] | NA [NA to NA] — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 8.93 [5.8 to 19.7]

8. Secondary Outcome: Tmax of Ezetimibe and Metabolite in Breast Milk
Description: Tmax of Ezetimibe and EZE-glucuronide in Breast Milk were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Hours | 2.93 [2.8 to 6.0] | 5.88 [2.8 to 8.9]

9. Secondary Outcome: Area Under the Breast Milk Concentration-time Curve Over the 24-hour Collection Interval (AUC24h) of Bempedoic Acid and Metabolites in Breast Milk
Description: AUC24h of ETC-1002, ESP-15228, and ETC-1002-glucuronide in Breast Milk were analyzed for Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Hours*nanograms per milliliter | 1765.86 (40.88) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 1308.84 (56.24) | 1618.25 (39.67) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 1057.69 (43.21)

10. Secondary Outcome: AUC24h of Ezetimibe and Metabolite in Breast Milk
Description: AUC24h of Ezetimibe and EZE-glucuronide in Breast Milk were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Hours*nanograms per milliliter | 7.79 (38.29) | 41.09 (66.10)

11. Secondary Outcome: Average Concentration (Cavg) of Bempedoic Acid and Metabolites in Breast Milk
Description: Cavg (defined as AUC24h/24h) of ETC-1002, ESP-15228, and ETC-1002-glucuronide in Breast Milk were analyzed for Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Nanograms per milliliter | 74.181 (40.75) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 54.982 (55.98) | 67.848 (39.77) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 44.346 (43.42)

12. Secondary Outcome: Cavg of Ezetimibe and Metabolite in Breast Milk
Description: Cavg of Ezetimibe and EZE-glucuronide in Breast Milk were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 0.327 (38.41) | 1.723 (66.03)

13. Secondary Outcome: Trough Concentration (Ctrough) of Bempedoic Acid and Metabolites in Breast Milk
Description: Ctrough_milk of ETC-1002, ESP-15228, and ETC-1002-glucuronide were analyzed for Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Nanograms per milliliter | 50.58 (47.59) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 45.55 (62.72) | 58.60 (53.36) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 39.32 (51.81)

14. Secondary Outcome: Ctrough of Ezetimibe and Metabolite in Breast Milk
Description: Ctrough_milk of Ezetimibe and EZE-glucuronide were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 0.25 (38.66) | 1.33 (82.37)

15. Secondary Outcome: Ctrough of Bempedoic Acid and Metabolites in Plasma
Description: Ctrough_plasma of ETC-1002, ESP-15228, and ETC-1002-glucuronide were analyzed for Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 8
Nanograms per milliliter | 10025.6 (25.46) | 1862.4 (34.04) | 4904.9 (35.65) | 9665.9 (37.95) | 1641.8 (20.78) | 4984.7 (35.65)

16. Secondary Outcome: Ctrough of Ezetimibe and Metabolite in Plasma
Description: Ctrough_plasma of Ezetimibe and EZE-glucuronide were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Nanograms per milliliter | 2.29 (69.37) | 35.76 (77.54)

17. Secondary Outcome: Ctrough_milk/Ctrough_plasma (M/P Ratio) of Bempedoic Acid and Metabolites
Description: M/P Ratio of ETC-1002, ESP-15228, and ETC-1002-glucuronide were analyzed for Bempedoic Acid arm and FCDP arm respectively.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set. Only those participants with data available at specified time points has been presented.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | ETC-1002 | ESP-15228 | ETC-1002-Glucuronide | ETC-1002 (FCDP) | ESP-15228 (FCDP) | ETC-1002-Glucuronide (FCDP)
Number analyzed (Participants) | 8 | 1 | 8 | 8 | 1 | 8
Ratio | 0.005 (25.35) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 0.009 (29.05) | 0.006 (59.39) | NA (NA) — Not applicable (NA) due to 7 out of 8 participants had ESP-15228 concentration below the lower limit of quantification (BLQ) (<20.0) at all nominal timepoints. | 0.008 (63.91)

18. Secondary Outcome: M/P Ratio of Ezetimibe and Metabolite
Description: M/P Ratio of Ezetimibe and EZE-glucuronide were analyzed for FCDP arm only.
Time Frame: 24 hours post Day 6 dose administration
Population: Pharmacokinetic Analysis Set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Ezetimibe | EZE-Glucuronide
Number analyzed (Participants) | 8 | 8
Ratio | 0.108 (62.21) | 0.037 (81.68)

ADVERSE EVENTS:
Time Frame: Up to Day 43
Description: Treatment emergent adverse events and serious adverse events were collected in Full Analysis Set.
Groups:
- Bempedoic Acid / Ezetimibe FCDP: Participants received bempedoic acid 180 mg/ezetimibe 10 mg FCDP oral tablets for 6 days
Arm/Group | Bempedoic Acid | Bempedoic Acid / Ezetimibe FCDP
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 3/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bempedoic Acid (N=8) | Bempedoic Acid / Ezetimibe FCDP (N=8)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 2
Rhinitis (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Principal Investigator plans to publish information from the study, a copy of the manuscript should be provided to the Sponsor for review before submission for publication or presentation. The Sponsor may request that that publication be withheld.

DOCUMENTS (2):
  • Study Protocol (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT06021951/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT06021951/SAP_001.pdf